CLINICAL TRIAL: NCT01306045
Title: Pilot Trial of Molecular Profiling and Targeted Therapy for Advanced Non-Small Cell Lung Cancer, Small Cell Lung Cancer, and Thymic Malignancies
Brief Title: Molecular Profiling and Targeted Therapy for Advanced Non-Small Cell Lung Cancer, Small Cell Lung Cancer, and Thymic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Arun Rajan, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110096; 11-C-0096
Record Dates: First submitted 2011-02-26; First posted 2011-03-01 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell Lung; Carcinoma, Thymic
Keywords: AZD6244; MK-2206; Lapatinib; Erlotinib; Sunitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Thymoma | interventions — AZD 6244; MK 2206; Lapatinib; Erlotinib Hydrochloride; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- A/ Erlotinib (Active Comparator): Arm A - Erlotinib 150 mg by mouth (PO) every morning (QAM)
  Interventions: Drug: Erlotinib; Procedure: Molecular Profiling
- B/ AZD6244 (Active Comparator): AZD6244 Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours
  Interventions: Drug: AZD6244; Procedure: Molecular Profiling
- C/ MK-2206 (Active Comparator): MK-2206 200 mg by mouth (PO) every (Q) Week
  Interventions: Drug: MK-2206; Procedure: Molecular Profiling
- D/ Lapatinib (Active Comparator): Lapatinib 1500 mg by mouth (PO) every day (QD)
  Interventions: Drug: Lapatinib; Procedure: Molecular Profiling
- E/Sunitinib (Active Comparator): Sunitinib 50 mg by mouth (PO) on days 1-28
  Interventions: Drug: Sunitinib; Procedure: Molecular Profiling
- F/ Not Otherwise Specified (NOS) (Other): Participants who do not meet the eligibility criteria for enrollment
  Interventions: Procedure: Molecular Profiling

INTERVENTIONS:
Drug: AZD6244 — Cycle = 21 days AZD6244 Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours
  Other Names: Selumetinib
  Arms: B/ AZD6244
Drug: MK-2206 — Cycle = 28 days MK-2206 200 mg by mouth (PO) every (Q) Week
  Arms: C/ MK-2206
Drug: Lapatinib — Cycle = 21 days Lapatinib 1500 mg by mouth (PO) every day (QD)
  Other Names: Tykerb
  Arms: D/ Lapatinib
Drug: Erlotinib — Cycle = 21 days Erlotinib 150 mg by mouth (PO) every morning (QAM)
  Other Names: Tarceva
  Arms: A/ Erlotinib
Drug: Sunitinib — Cycle = 42 days Sunitinib 50 mg by mouth (PO) on days 1-28
  Other Names: Sutent
  Arms: E/Sunitinib
Procedure: Molecular Profiling — Molecular profiling of tumor tissue. Not Otherwise Specified (NOS) arm. Participants who do not meet the eligibility criteria for enrollment or who meet eligibility criteria for a particular arm but can't be enrolled

SUMMARY:
Background:

- The current standard of care for advanced lung cancer and cancers of the thymus consists primarily of chemotherapy treatment. The drugs used for chemotherapy depend on the classification of the cancer in different categories that are based on the appearance of the cancer in the microscope. Though this approach has been proved to be useful in some ways, the survival rates of individuals with lung cancer and cancers of the thymus are still very poor. Recent research has shown that several genetic abnormalities play an important role in the development and growth of lung cancer and cancers of the thymus, and that it is possible to improve treatment success rates with drugs that specifically target some of the abnormal genes. Researchers are interested in determining whether it is possible to analyze the genes of patients with lung cancer and cancers of the thymus in order to provide personalized treatment with drugs that target the specific gene abnormalities.

Objectives:

- To evaluate the effectiveness of genetic analysis in determining targeted therapy for individuals with advanced non-small cell lung cancer, small cell lung cancer, and thymic cancer.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with either lung cancer or a cancer of the thymus that is not considered to be curable with the use of surgery or radiation therapy.

Design:

* Participants will be screened with a full medical history and physical examination, blood and urine tests, and tumor imaging studies. Participants will have a tumor biopsy or provide previously collected tumor tissue for study.
* Based on the results of the tumor biopsy study, participants will be separated into different treatment groups:
* Participants with epidermal growth factor receptor (EGFR) gene mutation will receive a drug called erlotinib, which inhibits a protein called EGFR that is thought to be a key factor in the development and progression of some cancers.
* Participants with Kirsten rat sarcoma virus (KRAS), proto-oncogene B-Raf (BRAF), Harvey Rat sarcoma virus (HRAS), or NRAF gene mutations will receive a drug called AZD6244, which inhibits a protein called methyl ethyl ketone (MEK) that is thought to be a key factor in the development and progression of some cancers.
* Participants with phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA), protein kinase B (AKT), or phosphatase and tensin homolog (PTEN) gene mutations will receive a drug called MK-2206, which inhibits a protein called AKT that is thought to be a key factor in the development and progression of some cancers.
* Participants with KIT or platelet-derived growth factor receptor A, (PDGFRA) gene mutations will receive a drug called sunitinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers, including kidney cancer.
* Participants who have -erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 (ERBB2) gene mutation or amplification will receive a drug called lapatinib, which inhibits some proteins that are thought to be key factors in the development and progression of some cancers, including breast cancer.
* Participants who do not have any of the genetic abnormalities described above will be offered different options for treatment, including standard of care chemotherapy or treatment with investigational agents in a different research protocol.
* After 6 weeks of treatment, participants will have imaging studies to evaluate the status of their cancer. Treatment will continue as long as participants tolerate the drugs, and the disease does not progress.
* Participants who benefit from the first treatment but eventually develop resistance and progression of their cancer will be offered the chance to have a second tumor biopsy and undergo a different treatment for their cancer.

DETAILED DESCRIPTION:
BACKGROUND:

* A better understanding of the genetic make-up of the individual tumor may offer potentially improved therapies. This approach may also give rapid access to response data in patients with sometimes rare genetic abnormalities.
* In addition, it will allow us to test targeted therapies in a select population of patients that is more likely to have a favorable response based on their molecular profile and the specific mechanism of action of the drug being tested.
* This approach will also speed up drug development and potentially approval and rescue an otherwise ineffective drug candidate for the specific subgroup that can benefit.

Primary Objectives:

* To determine the feasibility of the use of tumors molecular profiling and targeted therapies in the treatment of advanced stage non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC) and thymic malignancies.
* To estimate the response rate of molecular profile directed treatments in NSCLC, SCLC and thymic malignancies patients.

ELIGIBILITY:

* Patients with histologically confirmed advanced lung cancer or thymic malignancies for whom surgical resection with curative intent is not feasible.
* Patients must either have biopsiable disease and be willing to undergo biopsy for molecular profiling or have paraffin embedded tissue blocks suitable for molecular profiling analysis.
* Individuals are eligible for epidermal growth factor receptor (EGFR) germline mutation testing if they have:
* a personal history of invasive lung cancer or one of the pre-invasive histologies associated with the development of lung cancer and more than two affected family members with invasive lung cancer or one of the pre-invasive histologies associated with the development of lung cancer,

OR

* a first-degree relative with a known EGFR germline mutation (EGFR exon 20 T790M, exon 21 V843I, exon 21 R831C and exon 20 R776G).

DESIGN:

* All patients will have their tumors undergo molecular profiling. Based on these results and on other eligibility criteria, the patients will be offered enrollment into different targeted therapy arms.
* At the NCI site only, individuals eligible for EGFR germline mutation will undergo testing for germline mutations affecting the EGFR gene; if a mutation is detected, their first-degree relatives would be invited to undergo testing for the index germline mutation found in the proband and appropriate follow-up on trial.
* Effective with Amendment I, the participating site, Oregon Health and Science University (OHSU), will discontinue new enrollments and data entry for existing patients on the Not Other Specified (NOS) arm on this protocol in favor of the OHSU protocol L8639, Personalized Cancer Medicine Registry. The data from these patients will be included with the data from 11-C-0096 (8639) National Cancer Institute (NCI) patients at the time of publication. Any OHSU patients who are eligible for a treatment arm will continue to be enrolled and followed per protocol.

ELIGIBILITY:
* ELIGIBILITY CRITERIA FOR INITIAL ENROLLMENT:
* Patients with histologically confirmed advanced Non-Small Cell Lung Cancer, (NSCLC), Small Cell Lung Cancer (SCLC) and thymic malignancies for whom surgical resection or multimodality therapy with curative intent is not feasible. For patients with Stage III NSCLC, who can be encompassed by a radiation port, definitive radiation therapy (XRT) should have been performed first when possible.
* Individuals who meet the eligibility criteria for epidermal growth factor receptor (EGFR) germline mutation testing but who do not have advanced cancer as defined in 3.1.1 may enroll for EGFR germline mutation testing only and will not be eligible for the treatment or NOS arms.
* Patients with advanced cancer must meet one of the following criteria (does not apply to first degree relatives or individuals with pre-invasive histology enrolling only for EGFR germline mutation testing):

  * Patients must have biopsiable disease and be willing to undergo biopsy for molecular profiling

OR

-Patients must have enough and adequate archival material from a previous biopsy to perform molecular profiling analyses. The adequacy of the material provided will be determined by the principal investigator in conjunction with the laboratories performing the molecular profiling analyses

OR

* Patients must have previously undergone a successful molecular profiling of their tumor with mutation analysis of the genes described in section 5.2, as part of this protocol (crossover patients) or other molecular profiling protocols such as the Lung Cancer Mutation Consortium protocol among others.
* Age greater than or equal to18 years.

EXCLUSION CRITERIA:

1. Patients who have had major surgery, chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
2. Patients may not be receiving any other investigational agents or other medications for the treatment of their malignancy.
3. Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 1 week after the end of brain radiation may be enrolled to undergo molecular profiling at the discretion of the principal investigator. In addition, brain metastatic disease should be stable for at least 4 weeks, before the patients can be enrolled in any of the experimental treatment arms.
4. Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain tablets are excluded.
5. Any uncontrolled medical illness that precludes the patient from undergoing a biopsy for molecular profiling and/or receiving treatment under one of the experimental arms of the study should be excluded. These conditions include but are not limited to:

   * Ongoing or uncontrolled, symptomatic congestive heart failure (Class III or IV as defined by the New York Heart Association (NYHA) functional classification system (see Appendix D).
   * Uncontrolled hypertension
   * Unstable angina pectoris
   * Cardiac arrhythmia
   * Uncontrolled diabetes
   * Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients with corrected QT interval (QTc) prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities are excluded.
7. Caution should be used if patients are required to use a concomitant medication that can prolong the Q wave T wave (QT) interval and efforts should be made to switch to a different medication before the patient begins treatment under an experimental arm. See Appendix E for a table of medications with the potential to prolong the QTc interval. A comprehensive list of agents with the potential to cause QTc prolongation can be found at: http://www.azcert.org/medical-pros/drug-lists/bycategory.cfm
8. The eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the Principal Investigator. (A list of potent Cytochrome P450 3A4 (CYP3A4) inducers or inhibitors can be found in Appendix F). Every effort should be made to switch patients taking such agents or substances to other medications before they begin treatment with one of the experimental drug included in this protocol, particularly patients with gliomas or brain metastases who are taking enzyme-inducing anticonvulsant agents. A comprehensive list of medications and substances known or with the potential to alter the pharmacokinetics of sunitinib through CYP3A4 is provided in Appendix F.
9. Patients with tumor amenable to potentially curative therapy as assessed by the investigator.
10. Pregnant women are excluded from this study because many of the Food and Drug Administration (FDA) approved agents and investigational agents in this trial have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated in this protocol. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study PI. Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Adjei AA, Cohen RB, Franklin W, Morris C, Wilson D, Molina JR, Hanson LJ, Gore L, Chow L, Leong S, Maloney L, Gordon G, Simmons H, Marlow A, Litwiler K, Brown S, Poch G, Kane K, Haney J, Eckhardt SG. Phase I pharmacokinetic and pharmacodynamic study of the oral, small-molecule mitogen-activated protein kinase kinase 1/2 inhibitor AZD6244 (ARRY-142886) in patients with advanced cancers. J Clin Oncol. 2008 May 1;26(13):2139-46. doi: 10.1200/JCO.2007.14.4956. Epub 2008 Apr 7. PMID 18390968
- [Background] Allen LF, Sebolt-Leopold J, Meyer MB. CI-1040 (PD184352), a targeted signal transduction inhibitor of MEK (MAPKK). Semin Oncol. 2003 Oct;30(5 Suppl 16):105-16. doi: 10.1053/j.seminoncol.2003.08.012. PMID 14613031
- [Background] Altomare DA, Testa JR. Perturbations of the AKT signaling pathway in human cancer. Oncogene. 2005 Nov 14;24(50):7455-64. doi: 10.1038/sj.onc.1209085. PMID 16288292
- [Derived] Thomas A, Chen Y, Steinberg SM, Luo J, Pack S, Raffeld M, Abdullaev Z, Alewine C, Rajan A, Giaccone G, Pastan I, Miettinen M, Hassan R. High mesothelin expression in advanced lung adenocarcinoma is associated with KRAS mutations and a poor prognosis. Oncotarget. 2015 May 10;6(13):11694-703. doi: 10.18632/oncotarget.3429. PMID 26028668
- [Derived] Lopez-Chavez A, Thomas A, Rajan A, Raffeld M, Morrow B, Kelly R, Carter CA, Guha U, Killian K, Lau CC, Abdullaev Z, Xi L, Pack S, Meltzer PS, Corless CL, Sandler A, Beadling C, Warrick A, Liewehr DJ, Steinberg SM, Berman A, Doyle A, Szabo E, Wang Y, Giaccone G. Molecular profiling and targeted therapy for advanced thoracic malignancies: a biomarker-derived, multiarm, multihistology phase II basket trial. J Clin Oncol. 2015 Mar 20;33(9):1000-7. doi: 10.1200/JCO.2014.58.2007. Epub 2015 Feb 9. PMID 25667274
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0096.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: CUSTOM (Molecular Profiling and Targeted Therapies in Advanced Thoracic Malignancies). For efficacy, analysis data has been separated by type of intervention for each type of malignancy, e.g., Non-Small Cell Lung Cancer (NSCLC) pts receiving erlotinib, selumetinib etc. since results depend on the type of drug being administered.
Groups:
- Participants With Non-Small Cell Lung Cancer: Participants with tumors harboring epidermal growth factor receptor (EGFR) mutations; received Erlotinib 150 mg by mouth (PO) every morning (QAM); Participants with tumors harboring Kirsten rat sarcoma virus (KRAS), Harvey Rat sarcoma virus (HRAS), Neuroblastoma-RAS (NRAS), or proto-oncogene B-Raf (BRAF) mutations; received Selumetinib Sulfate (AZD6244) 75 mg by mouth (PO) every (Q) 12 Hours; Participants with tumors harboring phosphatase and tensin homolog (PTEN), protein kinase B (AKT) 1, or catalytic subunit alpha (PIK3CA) mutations; received MK-2206 200 mg by mouth (PO) every day (QD); Participants with tumors harboring -erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 (ERBB2) mutations or amplifications; received Lapatinib 1500 mg by mouth (PO) every day (QD); Participants with tumors harboring KIT or platelet-derived growth factor receptor A, (PDGFRA) mutations or amplifications; received Sunitinib 50 mg by mouth (PO) every day (QD).
- Participants With Small Cell Lung Cancer: Participants with tumors harboring epidermal growth factor receptor (EGFR) mutations; received Erlotinib 150 mg by mouth (PO) every morning (QAM); Participants with tumors harboring Kirsten rat sarcoma virus (KRAS),, Harvey Rat sarcoma virus (HRAS), Neuroblastoma-RAS (NRAS), or proto-oncogene B-Raf (BRAF) mutations; received Selumetinib Sulfate (AZD6244) 75 mg by mouth (PO) every (Q) 12 Hours; Participants with tumors harboring phosphatase and tensin homolog (PTEN), protein kinase B (AKT) 1, or catalytic subunit alpha (PIK3CA) mutations; received MK-2206 200 mg by mouth (PO) every day (QD); Participants with tumors harboring -erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 (ERBB2) mutations or amplifications; received Lapatinib 1500 mg by mouth (PO) every day (QD); Participants with tumors harboring KIT or P platelet-derived growth factor receptor A, (PDGFRA) mutations or amplifications; received Sunitinib 50 mg by mouth (PO) every day (QD).
- Participants With Thymic Malignancies: Participants with tumors harboring epidermal growth factor receptor (EGFR) mutations; received Erlotinib 150 mg by mouth (PO) every morning (QAM); Participants with tumors harboring Kirsten rat sarcoma virus (KRAS),, Harvey Rat sarcoma virus (HRAS), Neuroblastoma-RAS (NRAS), or proto-oncogene B-Raf (BRAF) mutations; received Selumetinib Sulfate (AZD6244) 75 mg by mouth (PO) every (Q) 12 Hours; Participants with tumors harboring phosphatase and tensin homolog (PTEN), protein kinase B (AKT) 1, or catalytic subunit alpha (PIK3CA) mutations; received MK-2206 200 mg by mouth (PO) every day (QD); Participants with tumors harboring -erb-b2 avian erythroblastic leukemia viral oncogene homolog 2 (ERBB2) mutations or amplifications; received Lapatinib 1500 mg by mouth (PO) every day (QD); Participants with tumors harboring KIT or platelet-derived growth factor receptor A, (PDGFRA) mutations or amplifications; received Sunitinib 50 mg by mouth (PO) every day (QD).
Period: Met General Eligibility Criteria
Arm/Group | Participants With Non-Small Cell Lung Cancer | Participants With Small Cell Lung Cancer | Participants With Thymic Malignancies
Started (647met eligibility criteria/underwent molecular profiling, 257 had 1 of the core mutations&45 enrolled in 1 of the treatment arms. 602 enrolled in Not Otherwise Specified Arm&received standard of care treatment or enrolled in other clinical trials&followed prospectively until death(312 with tumors-wild type or unknown for the mutation of interest, 212positive for 1 of the core mutations of interest but failed to enroll in treatment arms (screen failures)&78 with unsuccessful molecular profiling.) | 481 | 68 | 98
Had EGFR Mutations | 88 | 1 | 1
Had KRAS, HRAS, NRAS, or BRAF Mutations | 103 | 5 | 2
Had PTEN, Akt1, or PIK3CA Abnormalities | 22 | 7 | 2
Had ERBB2 Mutations or Amplifications | 13 | 1 | 1
Had KIT or PDGFRA Mutations or Amplifications | 5 | 1 | 5
Enrolled Onto Treatment Arm | 38 | 4 | 3
Completed | 288 | 57 | 90
Not Completed | 193 | 11 | 8
Not completed — Screen failures | 193 | 11 | 8
Period: Treatments Received
Arm/Group | Participants With Non-Small Cell Lung Cancer | Participants With Small Cell Lung Cancer | Participants With Thymic Malignancies
Started | 38 (Group could be evaluated for response and survival.) | 4 (Group could be evaluated for response and survival.) | 3 (Group could be evaluated for response and survival.)
Received Erlotinib: Arm 1, Arm 2, and Arm 3 Respectively. | 15 | 0 | 1
Received Selumetinib: Arm 4, Arm 5, and Arm 6 Respectively. | 9 | 1 | 0
Received MK2206: Arm 7, Arm 8, and Arm 9 Respectively. | 4 | 2 | 1
Received Lapatinib: Arm 10, Arm 11, and Arm 12 Respectively. | 6 | 1 | 0
Received Sunitinib: Arm 13, Arm 14, and Arm 15 Respectively. | 2 | 0 | 1
Completed | 36 | 4 | 3
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For demographics, data has been separated by type of malignancy only since disease characteristics are specific to each type of malignancy.
Groups:
- Non-Small Cell Lung Cancer (NSCLC): NSCLC participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
- Small Cell Lung Cancer (SCLC): SCLC participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
- Thymic Malignancies: Thymic malignancies participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
- Total: Total of all reporting groups
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies | Total
Number analyzed (Participants) | 481 | 68 | 98 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.59 (11.41) | 60.75 (9.75) | 53.79 (14.22) | 61.06 (12.11)
Age, Customized [Count of Participants; unit: Participants]
  Age 18-39 | 13 | 0 | 17 | 30
  Age 40-64 | 253 | 43 | 55 | 351
  Age >65 | 215 | 25 | 26 | 266
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 33 | 48 | 330
  Male | 232 | 35 | 50 | 317
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 384 | 60 | 76 | 520
  Black or African American | 39 | 2 | 9 | 50
  Asian | 42 | 4 | 10 | 56
  Other | 8 | 1 | 2 | 11
  Hispanic | 9 | 1 | 1 | 11
  Non-Hispanic | 472 | 67 | 97 | 636
Region of Enrollment [Number; unit: participants]
  United States | 481 | 68 | 98 | 647
Eastern Cooperative Oncology (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  ECOG 2 is in bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities.
  ECOG 3 is in bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  ECOG 4 is 100% bedridden.
  Participants
    0 | 75 | 7 | 13 | 95
    1 | 322 | 43 | 77 | 442
    2 | 64 | 12 | 7 | 83
    3-4 | 20 | 6 | 1 | 27
Histologic Feature of Tumor [Count of Participants; unit: Participants] — *Participants included in the SCLC category (n=68) included 65 participants with a clearly histologically define SCLC and 3 participants (other) whose tumors were classified as lung neuroendocrine tumor.
  Participants
    Adenocarcinoma | 363 | 0 | 0 | 363
    Squamous cell carcinoma | 64 | 0 | 0 | 64
    Small cell* | 0 | 65 | 0 | 65
    Thymoma | 0 | 0 | 41 | 41
    Thymic carcinoma | 0 | 0 | 48 | 48
    Other | 54 | 3 | 9 | 66
Smoking History [Count of Participants; unit: Participants]
  Never-smokers | 148 | 5 | NA — Total not calculated because data are not available (NA) in one or more arms. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Current or former smokers | 333 | 63 | NA — Total not calculated because data are not available (NA) in one or more arms. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Enrolled Participants Testing Positive for Genomic Abnormality
Description: To determine the feasibility of the use of tumor molecular profiling and targeted therapies in the treatment of Non-Small Cell Lung Cancer (NSCLC), Small Cell Lung Cancer (SCLC), and Thymic Malignancies, the trial will be evaluated by determining the percentage of enrolled participants with a genomic abnormality. Identifying molecular profiles may help identify new targeted treatments for cancer.
Time Frame: 1 year and 11 months
Population: For tolerability, data has been separated by type of malignancy since the information being conveyed represents overall tolerability in participants with a given malignancy.
Measure: Number; unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies
Number analyzed (Participants) | 481 | 68 | 98
percentage of participants
  Tumor protein p53 (TP53): number analyzed (Participants) | 284 | 43 | 98
  Tumor protein p53 (TP53) | 28.5 | 44.2 | 0
  Kirsten rat sarcoma virus (KRAS): number analyzed (Participants) | 366 | 49 | 92
  Kirsten rat sarcoma virus (KRAS) | 24.9 | 4.1 | 0
  Epidermal growth factor receptor (EGFR): number analyzed (Participants) | 398 | 51 | 92
  Epidermal growth factor receptor (EGFR) | 22.1 | 2.0 | 1
  PDGFRA amplifications: number analyzed (Participants) | 39 | 0 | 6
  PDGFRA amplifications | 12.8 |  | 0
  phosphoinositide 3-kinase (PIK3)CA amplifications: number analyzed (Participants) | 18 | 0 | 0
  phosphoinositide 3-kinase (PIK3)CA amplifications | 11.1 |  |
  Anaplastic lymphoma kinase (ALK) trans: number analyzed (Participants) | 335 | 0 | 86
  Anaplastic lymphoma kinase (ALK) trans | 8.7 |  | 0
  Discoidin Domain Receptor 2 (DDR2): number analyzed (Participants) | 15 | 0 | 0
  Discoidin Domain Receptor 2 (DDR2) | 6.7 |  |
  Phosphatidylinositol 3-kinase (PIK3R2): number analyzed (Participants) | 15 | 0 | 0
  Phosphatidylinositol 3-kinase (PIK3R2) | 6.7 |  |
  Protein Tyrosine Phosphatase Receptor Type D (PTPRD): number analyzed (Participants) | 15 | 0 | 0
  Protein Tyrosine Phosphatase Receptor Type D (PTPRD) | 6.7 |  |
  Serine/threonine kinase 11 (STK11): number analyzed (Participants) | 165 | 0 | 0
  Serine/threonine kinase 11 (STK11) | 5.5 |  |
  Retinoblastoma 1 (RB1): number analyzed (Participants) | 165 | 15 | 0
  Retinoblastoma 1 (RB1) | 4.8 | 33.3 |
  SWI/SNF Related, Matrix Associated Actin Dependent Regulator Of ChromatinSubfamilyA Member4(SMARCA4): number analyzed (Participants) | 165 | 0 | 0
  SWI/SNF Related, Matrix Associated Actin Dependent Regulator Of ChromatinSubfamilyA Member4(SMARCA4) | 4.8 |  |
  Cyclin-Dependent Kinase Inhibitor 2A (CDKN2A): number analyzed (Participants) | 180 | 0 | 0
  Cyclin-Dependent Kinase Inhibitor 2A (CDKN2A) | 4.4 |  |
  Phosphatase and tensin homolog (PTEN): number analyzed (Participants) | 181 | 21 | 1
  Phosphatase and tensin homolog (PTEN) | 4.4 | 9.5 | 0
  hosphatidylinositol 3-kinase (PIK3CA): number analyzed (Participants) | 285 | 47 | 64
  hosphatidylinositol 3-kinase (PIK3CA) | 3.9 | 8.5 | 2
  Catenin Beta 1 (CTNNB1): number analyzed (Participants) | 268 | 0 | 0
  Catenin Beta 1 (CTNNB1) | 3.4 |  |
  Neurofibromatosis type 1 (NF1): number analyzed (Participants) | 165 | 15 | 0
  Neurofibromatosis type 1 (NF1) | 3.0 | 6.7 |
  esenchymal-epithelial transition factor (MET): number analyzed (Participants) | 268 | 38 | 0
  esenchymal-epithelial transition factor (MET) | 3.0 | 2.6 |
  Human epidermal growth factor receptor 2 (HER2) amplifications: number analyzed (Participants) | 211 | 18 | 84
  Human epidermal growth factor receptor 2 (HER2) amplifications | 2.8 | 5.6 | 1
  Erb-B2 Receptor Tyrosine Kinase 2 (ERBB2): number analyzed (Participants) | 284 | 0 | 48
  Erb-B2 Receptor Tyrosine Kinase 2 (ERBB2) | 2.8 |  | 0
  Ataxia telangiectasia mutated (ATM): number analyzed (Participants) | 165 | 0 | 0
  Ataxia telangiectasia mutated (ATM) | 2.4 |  |
  Erb-B2 Receptor Tyrosine Kinase 4 (ERBB4): number analyzed (Participants) | 165 | 0 | 0
  Erb-B2 Receptor Tyrosine Kinase 4 (ERBB4) | 2.4 |  |
  B-Raf Proto-Oncogene, Serine/Threonine Kinase (BRAF): number analyzed (Participants) | 349 | 68 | 92
  B-Raf Proto-Oncogene, Serine/Threonine Kinase (BRAF) | 2.3 | 2.0 | 0
  Smoothened (SMO): number analyzed (Participants) | 104 | 0 | 0
  Smoothened (SMO) | 1.9 |  |
  Neurotrophic Receptor Tyrosine Kinase 3 (NTRK3): number analyzed (Participants) | 118 | 0 | 0
  Neurotrophic Receptor Tyrosine Kinase 3 (NTRK3) | 1.7 |  |
  Phosphoinositide-3-Kinase Regulatory Subunit 1 (PIK3R1): number analyzed (Participants) | 118 | 0 | 0
  Phosphoinositide-3-Kinase Regulatory Subunit 1 (PIK3R1) | 0.8 |  |
  neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS): number analyzed (Participants) | 284 | 46 | 64
  neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS) | 0.7 | 2.2 | 0
  Harvey Rat sarcoma virus (HRAS): number analyzed (Participants) | 285 | 43 | 7
  Harvey Rat sarcoma virus (HRAS) | 0.7 | 2.3 | 0
  Tet Methylcytosine Dioxygenase 2 (TET2): number analyzed (Participants) | 267 | 15 | 0
  Tet Methylcytosine Dioxygenase 2 (TET2) | 0.4 | 6.7 |
  AKT Serine/Threonine Kinase 1 (AKT1): number analyzed (Participants) | 283 | 45 | 64
  AKT Serine/Threonine Kinase 1 (AKT1) | 0.4 | 2.2 | 0
  Neurogenic locus notch homolog protein 1 (NOTCH1): number analyzed (Participants) | 0 | 21 | 0
  Neurogenic locus notch homolog protein 1 (NOTCH1) |  | 4.8 |
  KIT Proto-Oncogene, Receptor Tyrosine Kinase (KIT): number analyzed (Participants) | 0 | 38 | 7
  KIT Proto-Oncogene, Receptor Tyrosine Kinase (KIT) |  | 2.6 | 0

2. Primary Outcome: Number of Evaluable Participants With a Response Based on Molecular Profile Directed Treatments in Non-Small Cell Lung Cancer, (NSCLC), Small Cell Lung Cancer (SCLC), and Thymic Malignancies
Description: Efficacy will be determined by assessing if participants who have treatment assigned on the basis of their molecular profiling results will exhibit reasonable response to the drug selected for their particular profile. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study Progressive Disease (PD) is At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 1 year and 13 months
Population: Overall number of participants analyzed represent the total number of participants for each tumor type evaluable for response (efficacy) across different treatment arms. For tolerability, data has been separated by type of malignancy since the information being conveyed represents overall tolerability in participants with a given malignancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies
Number analyzed (Participants) | 36 | 4 | 3
Participants
  Partial Response with Erlotinib: number analyzed (Participants) | 15 | 0 | 1
  Partial Response with Erlotinib | 9 |  | 0
  Stable Disease with Erlotinib: number analyzed (Participants) | 15 | 0 | 1
  Stable Disease with Erlotinib | 5 |  | 0
  Progressive Disease with Erlotinib: number analyzed (Participants) | 15 | 0 | 1
  Progressive Disease with Erlotinib | 1 |  | 1
  Partial Response to Lapatinib: number analyzed (Participants) | 6 | 1 | 0
  Partial Response to Lapatinib | 0 | 0 | 0
  Stable Disease with Lapatinib: number analyzed (Participants) | 6 | 1 | 0
  Stable Disease with Lapatinib | 4 | 1 |
  Progressive Disease with Lapatinib: number analyzed (Participants) | 6 | 1 | 0
  Progressive Disease with Lapatinib | 2 | 0 |
  Partial Response with Sunitinib: number analyzed (Participants) | 2 | 0 | 1
  Partial Response with Sunitinib | 0 |  | 0
  Stable Disease with Sunitinib: number analyzed (Participants) | 2 | 0 | 1
  Stable Disease with Sunitinib | 1 |  | 1
  Progressive Disease with Sunitinib: number analyzed (Participants) | 2 | 0 | 1
  Progressive Disease with Sunitinib | 1 |  | 0
  Partial Response with Selumetinib: number analyzed (Participants) | 9 | 1 | 0
  Partial Response with Selumetinib | 1 | 0 |
  Stable Disease with Selumetinib: number analyzed (Participants) | 9 | 1 | 0
  Stable Disease with Selumetinib | 4 | 0 |
  Progressive Disease with Selumetinib: number analyzed (Participants) | 9 | 1 | 0
  Progressive Disease with Selumetinib | 4 | 1 |
  Partial Response with MK2206: number analyzed (Participants) | 4 | 2 | 1
  Partial Response with MK2206 | 0 | 0 | 0
  Stable Disease with MK2206: number analyzed (Participants) | 4 | 2 | 1
  Stable Disease with MK2206 | 4 | 0 | 1
  Progressive Disease with MK2206: number analyzed (Participants) | 4 | 2 | 1
  Progressive Disease with MK2206 | 0 | 2 | 0

3. Primary Outcome: Percentage of Evaluable Participants Overall Response Rate (ORR) Based on the Drug Selected for Their Particular Profile
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).Partial Response (PD) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study Progressive Disease (PD) is At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 1 year and 13 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies
Number analyzed (Participants) | 36 | 4 | 3
percentage of participants
  Overall response rate to Erlotinib: number analyzed (Participants) | 15 | 0 | 1
  Overall response rate to Erlotinib | 60 [32.3 to 83.7] |  | 0 [0 to 0]
  Overall response rate to Lapatinib: number analyzed (Participants) | 6 | 1 | 0
  Overall response rate to Lapatinib | 0 [0 to 0] | 0 [0 to 0] |
  Overall response rate to Sunitinib: number analyzed (Participants) | 2 | 0 | 1
  Overall response rate to Sunitinib | 0 [0 to 0] |  | 0 [0 to 0]
  Overall response rate to Selumetinib: number analyzed (Participants) | 9 | 1 | 0
  Overall response rate to Selumetinib | 11 [0 to 48] | 0 [0 to 0] |
  Overall response rate to MK2206: number analyzed (Participants) | 4 | 2 | 1
  Overall response rate to MK2206 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Other Pre Specified Outcome: Frequency of Epidermal Growth Factor Receptor (EGFR) Germline Mutations in Families With High Susceptibility to Lung Cancer
Description: The frequency of EGFR germline mutations will be determined by enrolling participants from families with high susceptibility to lung cancer and their first-degree relatives (at the National Cancer Institute (NCI) site only). Individuals were tested for Epidermal Growth Factor Receptor (EGFR) Germline Mutations if they consented to participation in the study and had a personal history of invasive NSCLC or one of the pre-invasive histologies associated with the development of non-small cell lung cancer (NSCLC) and more than two affected family members with invasive NSCLC or one of the pre-invasive histologies associated with the development of NSCLC; OR a first-degree relative with a known EGFR germline mutation (EGFR threonine (T) with methionine (M) at position 790 of exon 20 (T790M), exon 21 V843I, exon 21 R831C and exon 20 R776G).
Time Frame: 5 years
Population: As pre-specified in the protocol, only the NSCLC group is reported here.
Measure: Number; unit: percentage of participants
Groups:
- Non-Small Cell Lung Cancer (NSCLC): Eligibility for this outcome measure was based on one or more of the following criteria: Personal history of invasive lung cancer or one of the pre-invasive histologies associated with the development of lung cancer [adenocarcinoma in situ (AIS), minimally invasive adenocarcinomas (MIA) or atypical adenomatous hyperplasia (AAH)] and more than two affected family members with invasive lung cancer or one of the pre-invasive histologies associated with the development of lung cancer; OR First-degree relatives of an individual enrolled in the study with a known EGFR germline mutation; OR Detection of de-novo (prior to any treatment with tyrosine kinase inhibitor (TKI) T790M mutation in the tumor specimen of a lung cancer patient; OR A family history of lung cancer not possibly related to smoking history, defined as at least one family member within the 3rd degree of consanguinity with lung cancer who was a never or oligo-smoker or at least two family members in either the maternal or paternal side with a history of lung cancer; OR Documented germline lung cancer associated mutation (such as EGFR T790M) tested elsewhere.
Arm/Group | Non-Small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 19
percentage of participants | 36.8

5. Other Pre Specified Outcome: Here is the Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 122 months and 25 days, 88 months and 16 days, and 126 months and 2 days for each group respectively.
Population: Serious and/or Non-Serious adverse events data was collected for 423/647 participants because the remainder did not undergo any study-related intervention because a new biopsy was not performed (archival tissue was used for molecular profiling) and/or the participant failed to enroll in one of the treatment arms. For tolerability, data has been separated by type of malignancy since the information being conveyed represents overall tolerability in participants with a given malignancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies
Number analyzed (Participants) | 310 | 22 | 91
Participants | 37 | 1 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 122 months and 25 days, 88 months and 16 days, and 126 months and 2 days for each group respectively.
Description: Data was collected for 423/647 participants(pts) because the remainder did not undergo any study-related intervention because a new biopsy wasn't performed(archival tissue was used for molecular profiling)and/or the pt failed to enroll in one of the treatment arms.All pts included in the mortality section. Data reported as an aggregate of events observed in pts with each tumor type who received any type of drug intervention (data is reported per tumor type and not per type of drug intervention).
Groups:
- Non-Small Cell Lung Cancer (NSCLC): NSCLC participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
  This protocol was designed to evaluate the feasibility of using tumor molecular profile and targeted therapies in the treatment of advanced thoracic malignancies. Assessment of adverse events (AEs) per therapeutic intervention was not an objective of this trial. Therefore, we have reported adverse events in aggregate form per histology and not as AEs per therapeutic intervention per histology.
- Small Cell Lung Cancer (SCLC): SCLC participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
  This protocol was designed to evaluate the feasibility of using tumor molecular profile and targeted therapies in the treatment of advanced thoracic malignancies. Assessment of adverse events (AEs) per therapeutic intervention was not an objective of this trial. Therefore, we have reported adverse events in aggregate form per histology and not as AEs per therapeutic intervention per histology.
- Thymic Malignancies: Thymic malignancies participants received Erlotinib 150 mg by mouth (PO) every morning (QAM), Selumetinib (AZD6244) Hydrogen Sulfate 75 mg by mouth (PO) every (Q) 12 Hours, MK-2206 200 mg by mouth (PO) every (Q) Week, Lapatinib 1500 mg by mouth (PO) every day (QD), and/or Sunitinib 50 mg by mouth (PO) on days 1-28.
  This protocol was designed to evaluate the feasibility of using tumor molecular profile and targeted therapies in the treatment of advanced thoracic malignancies. Assessment of adverse events (AEs) per therapeutic intervention was not an objective of this trial. Therefore, we have reported adverse events in aggregate form per histology and not as AEs per therapeutic intervention per histology.
Arm/Group | Non-Small Cell Lung Cancer (NSCLC) | Small Cell Lung Cancer (SCLC) | Thymic Malignancies
All-Cause Mortality (participants affected / at risk) | 467/481 | 68/68 | 88/98
Serious Adverse Events (participants affected / at risk) | 15/310 | 0/22 | 3/91
Other Adverse Events (participants affected / at risk) | 37/310 | 1/22 | 3/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Small Cell Lung Cancer (NSCLC) (N=310) | Small Cell Lung Cancer (SCLC) (N=22) | Thymic Malignancies (N=91)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 7 (7) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death during follow up (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignant Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Non-Small Cell Lung Cancer (NSCLC) (N=310) | Small Cell Lung Cancer (SCLC) (N=22) | Thymic Malignancies (N=91)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0)
Alanine aminotransferase increased (Investigations) | 7 (8) | 0 (0) | 0/0 (0)
Alkaline phosphatase increased (Investigations) | 6 (10) | 0 (0) | 0/0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0/0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0/0 (0)
Anemia (Blood and lymphatic system disorders) | 10 (17) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (8) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 3 (5) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Edema face (General disorders) | 4 (6) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 4 (7) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Periorbital edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Elongated Eyelashes (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (10) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Mouth ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Sensation of swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (16) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 13 (22) | 0 (0) | 3 (7)
Lymphocyte count increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 8 (10) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 4 (6) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (11) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (14) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Ichthyosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 3 (4) | 0 (0) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT01306045/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT01306045/ICF_001.pdf